CLINICAL TRIAL: NCT07283575
Title: ctDNA Methylation for Efficacy Assessment and Prognostic Prediction in Advanced Colorectal Cancer Treated With Radiotherapy Combined With or Without PD-1 Inhibitor: A Prospective Cohort Study (PROMET)
Brief Title: Using ctDNA Methylation to Monitor Metastatic Colorectal Cancer Treatment (PROMET)
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, MD, PhD, Fudan University
Other Study IDs: 2025-364-4513
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer ctDNA Surveillance
Keywords: Metastatic Colorectal Cancer(mCRC); Radiotherapy; Immunotherapy; ctDNA methylation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Newly diagnosed, histologically confirmed, recurrent or metastatic colorectal cancer, amenable to receive radiotherapy in combination with standard-of-care chemotherapy, with or without PD-1 inhibitors.
  Patients will receive dynamic monitoring of ctDNA + routine follow-up: ctDNA detection is performed at baseline, multiple predefined timepoints during treatment and follow-up for a period of 2 years. At the same time, participants will undergo routine imaging surveillance (CT/MRI) every three months.
  Interventions: Diagnostic Test: Plasma ctDNA methylation profiling

INTERVENTIONS:
Diagnostic Test: Plasma ctDNA methylation profiling — Plasma ctDNA methylation profiling was performed using an optimized single-tube multiplex mqMSP assay

SUMMARY:
Multi-center observational clinical study to evaluate the application value of ctDNA methylation monitoring in efficacy assessment and relapse prediction in patients diagnosed with recurrence or metastatic colorectal cancer receiving radiotherapy plus SOC with or without PD-1.

DETAILED DESCRIPTION:
This study will enroll patients with histologically confirmed, recurrent or metastatic colorectal cancer who are eligible to receive radiotherapy in combination with standard-of-care chemotherapy, with or without PD-1 inhibitors. The study will employ ctDNA methylation detection technology to quantitatively assess ctDNA methylation levels in patient plasma samples. Blood samples will be collected at baseline and at multiple predefined timepoints during treatment. In addition, participants will undergo standard imaging surveillance (CT/MRI) every three months. The study aims to correlate ctDNA dynamics with therapeutic response, time to recurrence, and survival outcomes. Ultimately, it seeks to evaluate the potential of ctDNA monitoring for predicting treatment efficacy and prognosis, and to explore its utility in guiding clinical management for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Histologically confirmed, recurrent or metastatic colorectal cancer;
3. Eligible to receive radiotherapy in combination with standard-of-care chemotherapy, with or without PD-1 inhibitors.
4. With expected survival of more than 6 months;
5. The subjects (or their legal representative / Guardian) must sign the informed consent form, indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study.

Exclusion Criteria:

1. Blood transfusion performed during operation or within 2 weeks before operation;
2. Pregnant or lactating women who have fertility and do not take adequate contraceptive measures;
3. Have a history of other malignant tumors within 5 years, except cured cervical carcinoma in situ or non melanoma skin cancer;
4. Primary brain tumor or central nerve metastasis is not under control, with obvious intracranial hypertension or neuropsychiatric symptoms;
5. Patients with the following serious or uncontrollable diseases: severe heart disease, the condition is still unstable after treatment, including myocardial infarction, congestive heart failure, unstable angina pectoris, pericardial effusion with obvious symptoms or unstable arrhythmia within 6 months before enrollment; definite neuropathy or psychosis, including dementia or seizures; severe or uncontrolled infection; active disseminated intravascular coagulation and obvious bleeding tendency;
6. Significant impairment of important organ function;
7. Other conditions in which the investigator believes that the patient should not participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed, recurrent or metastatic colorectal cancer who are eligible to receive radiotherapy in combination with standard-of-care chemotherapy, with or without PD-1 inhibitors.
Sampling Method: Probability Sample
Enrollment: 497 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2028-10-10 (Estimated); Study Completion 2030-10-10 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2 years
  To investigate ctDNA-based disease-free survival (ctDNA-DFS), CT-based disease-free survival (CT-DFS), and the difference between ctDNA-DFS and CT-DFS (△-DFS).

SECONDARY OUTCOMES:
OS | up to 5 year
  To exam whether 3- and 5-year overall survival (OS) with ctDNA-guided surveillance is comparable to that achieved with standard CT-based monitoring.
Patient-reported outcomes (quality of life) | up to 5 year
  To assess patient-reported outcomes-quality of life (EORTC QLQ-C30)-in those receiving ctDNA-guided versus standard surveillance.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No